CLINICAL TRIAL: NCT06934577
Title: Michigan Screening and Intervention for Glaucoma and Eye Health Through Telemedicine- SIGHT 2: A Pragmatic Randomized Trial
Brief Title: Michigan Screening and Intervention for Glaucoma and Eye Health Through Telemedicine (SIGHT) 2
Acronym: SIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paula Anne Newman-Casey, Professor of Ophthalmology and Visual Sciences, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00267229; 1 U01DP006826-01-00 (Other: Centers for Disease Control and Prevention); 1U01DP006826-01 (NIH)
Record Dates: First submitted 2025-04-10; First posted 2025-04-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Eye Diseases; Visual Impairment; Glaucoma
Keywords: Eye disease screening; Glaucoma detection
MeSH Terms: conditions — Eye Diseases; Vision Disorders; Glaucoma

STUDY DESIGN:
Intervention Model Description: Participants meeting inclusion criteria who are 18 years of age or older will be randomized to either 1) control group: standard optometric examination or 2) intervention group: technology-enhanced eye disease screening protocol. Randomization will be stratified by disease risk in two strata: 1) those with and without diabetes, and 2) those < age 40 and those ≥ age 40. After stratification, participants will be block randomized to the control or intervention arm.
Who Masked: Outcomes Assessor
Masking Description: The statistician assessing the main outcome measure will be masked. A second statistician, not masked to treatment allocation, will tabulate weekly reports of adverse events by treatment group for review by the medical monitor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control, standard optometric examination (Experimental): Participants will receive usual care with an optometrist with a biomicroscopic exam at the Federally Qualified Health Center to identify eye disease.
  Interventions: Other: Standard optometric examination; Other: Technology enhanced eye disease detection protocol
- Intervention, technology enhanced eye disease detection protocol (Experimental): Participants will receive a technology enhanced eye disease detection protocol from ophthalmic technicians that includes measurements of visual function such as visual acuity, refraction, intraocular pressure, pachymetry, external eye and fundus photography, and optical coherence tomography of the macula and retinal nerve fiber layer. The optometrist at the Federally. Qualified Health Center will then use a protocol to grade the testing and identify eye disease. The results of the grading will inform whether the person receives a brief appointment with the optometrist (if no disease is detected) or an in-depth appointment with the optometrist (if there is disease detected).
  Interventions: Other: Standard optometric examination; Other: Technology enhanced eye disease detection protocol

INTERVENTIONS:
Other: Standard optometric examination — Participants will see the optometrist at the Federally Qualified Health Center. The guidelines define usual care as: an in-person comprehensive eye examination with assessment of patient history, visual acuity, pupil examination, ocular motility and alignment, intraocular pressure, and biomicroscopy with additional tests, as appropriate. A glasses prescription will be given to the participant if needed. Participants will complete surveys at baseline before their eye exam and 6 weeks after the eye exam.
Other: Technology enhanced eye disease detection protocol — Participants will receive a technology enhanced eye disease detection protocol from ophthalmic technicians that includes measurements of visual function such as visual acuity, refraction, intraocular pressure, pachymetry, external eye and fundus photography, and optical coherence tomography of the macula and retinal nerve fiber layer. The optometrist at the Federally. Qualified Health Center will then use a protocol to grade the testing and identify eye disease. The results of the grading will inform whether the person receives a brief appointment with the optometrist (no disease detected) or an in-depth appointment with the optometrist (disease detected). During the first visit, participants receive care navigation support to purchase low-cost glasses from an on-line retailer. When participants return for the optometrist exam, glasses will be fit. Participants will receive care navigation support to attend any recommended specialty follow-up appointments.

SUMMARY:
To compare eye disease detection rates at a Federally Qualified Health Center between a technology-enhanced protocol and standard optometric clinical examination for three of the leading causes of blindness: glaucoma, diabetic retinopathy, and visually significant cataract.

ELIGIBILITY:
Inclusion Criteria:

• Speak English, Spanish, Arabic, Chinese, French, Hindi, Finnish, Albanian, Russian or Tagalog

Exclusion Criteria:

* significant eye pain
* sudden decrease in vision within one week
* binocular diplopia
* cognitive impairment
* pregnancy
* previously declined participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Rate of vision threatening eye disease (glaucoma/suspected glaucoma, visually significant cataract, diabetic retinopathy) | Visit 1(day 1)
Rate of glaucoma/suspected glaucoma | Visit 1 (Day 1)
Rate of visually significant cataract | Visit 1(day 1)
  Visually significant cataract is defined as presence of cataract with best corrected visual acuity ≤ 20/40 in the absence of other pathology.
Rate of diabetic retinopathy | Visit 1(day 1)

SECONDARY OUTCOMES:
Visual Function | 6 weeks
  The Visual Function Questionnaire (VFQ-9) is a 9-item survey that measures vision related quality-of-life and is scored from 0-100, where 100 represents the best visual function and vision-related quality-of-life.
Rate of disease in second allocation | 6 weeks
  Rate of glaucoma/glaucoma suspect in second allocation

CONTACTS AND LOCATIONS:
Overall Officials: Paula Anne Newman-Casey, MD, Principal Investigator — University of Michigan
Locations (1):
- Hamilton Optometry Clinic, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No